CLINICAL TRIAL: NCT05821257
Title: Arm Swing During Walking in Early Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gokce Leblebici, Physiotherapist, Istanbul Medeniyet University
Other Study IDs: IstanbulUC_MStation_armswing
Record Dates: First submitted 2023-03-27; First posted 2023-04-20 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis; Upper Extremity Problem; Gait Disorders, Neurologic
Keywords: arm swing, multiple sclerosis, gait, foot pressure analysis
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Multiple Sclerosis: Arm swing evaluation and functional tests will be tested in this group.
  Interventions: Other: Evaluation of the arm swing during gait; Other: Functional Tests
- Healthy Controls: Arm swing evaluation will be tested in this group.
  Interventions: Other: Evaluation of the arm swing during gait

INTERVENTIONS:
Other: Evaluation of the arm swing during gait — Evaluation of the arm swing during gait: The difference between the maximum flexion and extension of the shoulder is the arm swing amplitude during walking. The arm swing amplitude will be evaluated 2-dimensionally with the help of the Kinovea video player.
  Other Names: Arm swing during walking
Other: Functional Tests — To understand the changes in functional mobility, Two Minute Walk Test (2MWT), Timed Up and Go (TUG) and Timed 25Foot Walk Test (T25FW) were conducted.
  Other Names: Two Minute Walk Test (2MWT), Timed Up and Go (TUG) and Timed 25Foot Walk Test (T25FW)
  Groups: Early Multiple Sclerosis

SUMMARY:
Multiple sclerosis (MS) is the most common central nervous system inflammatory demyelinating disease which causes motor and sensory deficits, cerebellar symptoms, and balance problems. Due to these symptoms, gait abnormalities are common in MS, even in patients with low degrees of impairment. The upper limb has an important role on postural control and gait stability. Affected arm swing movement and asymmetry during gait are common in neurological disorders such as Parkinson's disease (PD) even in early stages of the disease and arm swing treatment has been acknowledged to enhance gait and normalize arm swing in individuals with PD.

The presence of arm swing changes during walking in MS patients, similar to PD, especially in the early period, may be an indicator of balance problems, this was, however, not investigated as such. Therefore, the aim of the current study is to assess the arm swing during gait in people with MS shortly after their diagnosis in early MS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with MS in the last 30 days,
* Patients who were recovered from their symptoms and were clinically stable

Exclusion Criteria:

* Patients who had an acute medical illness in the past 6 months, any other neurological and psychiatric diseases
* Patients who had any orthopedic, rheumatologic, or vestibular conditions that affect walking
* Patients who had exacerbations between the first and second evaluations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eighteen MS outpatients from a hospital and 10 healthy controls were included. The patients who were diagnosed with MS in the last 30 days, were recovered from their symptoms and were clinically stable were included.
  Patients who had an acute medical illness in the past 6 months, any other neurological and psychiatric diseases, and any orthopedic, rheumatologic, or vestibular conditions that affect walking were excluded. The patients who had exacerbations between the first and second evaluations (three months after the first evaluation) were excluded.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Arm swing amplitude-shoulder degrees in flexion-extension direction | 3 months after the baseline
  The difference between the maximum flexion and extension of the shoulder will be calculated with Kinovea video player.
Arm swing amplitude-elbow degrees in flexion-extension direction | 3 months after the baseline
  The difference between the maximum flexion and extension of the shoulder will be calculated with Kinovea video player.
Arm swing amplitude-overall degrees in flexion-extension direction | 3 months after the baseline
  The difference between the maximum flexion and extension of the shoulder will be calculated with Kinovea video player.
Step-speed | 3 months after the baseline
  The stepping task required patients to walk back and forth for 2 minutes over a three meters walkway which was set up with the FreeMed foot pressure analysis system (Sensor Medica, Guidonia Montecelio). Step speed outcome was collected from foot pressure analysis system.
Two Minute Walk Test (2MWT) | 3 months after the baseline
  It is a measure of self-paced walking ability and functional capacity. The person is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured.
Timed Up and Go (TUG) | 3 months after the baseline
  To determine fall risk and measure the progress of balance, sit to stand and walking.It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees.
Timed 25Foot Walk Test (T25FW) | 3 months after the baseline
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Kalinowska-Lyszczarz A, Guo Y, Lucchinetti CF. Update on pathology of central nervous system inflammatory demyelinating diseases. Neurol Neurochir Pol. 2022;56(3):201-209. doi: 10.5603/PJNNS.a2022.0046. Epub 2022 Jun 27. PMID 35758517
- [Background] Morel E, Allali G, Laidet M, Assal F, Lalive PH, Armand S. Gait Profile Score in multiple sclerosis patients with low disability. Gait Posture. 2017 Jan;51:169-173. doi: 10.1016/j.gaitpost.2016.10.013. Epub 2016 Oct 18. PMID 27776271
- [Background] Meyns P, Bruijn SM, Duysens J. The how and why of arm swing during human walking. Gait Posture. 2013 Sep;38(4):555-62. doi: 10.1016/j.gaitpost.2013.02.006. Epub 2013 Mar 13. PMID 23489950
- [Background] Gholizadeh H, Hill A, Nantel J. The effect of various arm and walking conditions on postural dynamic stability when recovering from a trip perturbation. Gait Posture. 2020 Feb;76:284-289. doi: 10.1016/j.gaitpost.2019.11.010. Epub 2019 Dec 17. PMID 31884255
- [Background] Lewek MD, Poole R, Johnson J, Halawa O, Huang X. Arm swing magnitude and asymmetry during gait in the early stages of Parkinson's disease. Gait Posture. 2010 Feb;31(2):256-60. doi: 10.1016/j.gaitpost.2009.10.013. Epub 2009 Nov 27. PMID 19945285
- [Background] Koh SB, Park YM, Kim MJ, Kim WS. Influences of elbow, shoulder, trunk motion and temporospatial parameters on arm swing asymmetry of Parkinson's disease during walking. Hum Mov Sci. 2019 Dec;68:102527. doi: 10.1016/j.humov.2019.102527. Epub 2019 Nov 2. PMID 31689575
- [Background] Elsworth-Edelsten C, Bonnefoy-Mazure A, Laidet M, Armand S, Assal F, Lalive P, Allali G. Upper limb movement analysis during gait in multiple sclerosis patients. Hum Mov Sci. 2017 Aug;54:248-252. doi: 10.1016/j.humov.2017.05.014. Epub 2017 May 30. PMID 28575710
- [Background] Yoon J, Park J, Park K, Jo G, Kim H, Jang W, Kim JS, Youn J, Oh ES, Kim HT, Youm CH. The effects of additional arm weights on arm-swing magnitude and gait patterns in Parkinson's disease. Clin Neurophysiol. 2016 Jan;127(1):693-697. doi: 10.1016/j.clinph.2015.06.005. Epub 2015 Jun 15. PMID 26183756